CLINICAL TRIAL: NCT02831894
Title: The Role of Tapering Pace and Selected Traits on Hypnotic Discontinuation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-2891
Record Dates: First submitted 2016-05-13; First posted 2016-07-13 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Hypnotic Dependence Among Those With Insomnia
Keywords: insomnia; sedative hypnotics; hypnotic tapering
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0% Hypnotic Medication Taper (Sham Comparator): In this condition patients will be maintained on their baseline hypnotic medication dosage throughout a 20-week double-blinded tapering period.
  Interventions: Drug: 0% Hypnotic Medication Taper
- 25% Hypnotic Medication Taper (Active Comparator): In this condition patients will have their current hypnotic medication dosage reduced by 25% every 2 weeks throughout a 20-week double-blinded tapering period.
  Interventions: Drug: 25% Hypnotic Medication Taper
- 10% Hypnotic Medication Taper (Active Comparator): In this condition patients will have their current hypnotic medication dosage reduced by 10% every 2 weeks throughout a 20-week double-blinded tapering period.
  Interventions: Drug: 10% Hypnotic Medication Taper

INTERVENTIONS:
Drug: 0% Hypnotic Medication Taper — Participants will not have their soporific hypnotic medication dosage changed during a 20 week blinded tapering period
  Other Names: No Drug Taper
  Arms: 0% Hypnotic Medication Taper
Drug: 25% Hypnotic Medication Taper — Participants will have their soporific hypnotic medication dosage reduced by 25% every two weeks during a 20 week blinded tapering period.
  Other Names: Quarter Drug Taper
  Arms: 25% Hypnotic Medication Taper
Drug: 10% Hypnotic Medication Taper — Participants will have their soporific hypnotic medication dosage reduced by 10% every two weeks during a 20 week blinded tapering period.
  Other Names: Tenth Drug Taper
  Arms: 10% Hypnotic Medication Taper

SUMMARY:
Treatment seeking insomnia sufferers most often present in primary care venues where the first and usually only treatment is a prescription for a sedative hypnotic, typically a benzodiazepine or newer benzodiazepine receptor agonist, For some patients, short term or intermittent use provides satisfactory insomnia relief. However, more than 65 percent of individuals who are prescribed hypnotics use them for more than a year, and over 30 percent remain on these agents for more than five years. Whereas some patients may appreciate partial or full relief of insomnia symptoms with ongoing hypnotic use, continuous long-term use of these agents may not represent optimal therapy. Many insomnia patients who participate in non drug insomnia therapy such as as cognitive behavioral insomnia therapy or Cognitive Behavioral Therapy For Insomnia (CBTI) achieve sustained insomnia remission lon after a time limited course of treatment. However it is difficult for most long term hypnotic users to convert to a self management approach. Intervention that combine CBTI with a supervised medication tapering (SMT) have shown the greatest promise for achieving this outcome, but almost 50 percent of patients who receive this treatment either fail to discontinue hypnotics or resume them over time. Previous research provides only rudimentary understanding of how to help long term hypnotic users discontinue their sleep aids and successfully manage their insomnia with CBTI techniques. This R34 gathered key pilot data to address these limitations. Specifically this project compared the currently recommended tapering pace which is a 25 percent dose reduction every two weeks with a slower 10 percent dose reduction every two weeks. The study also conducted all tapering in double blinded fashion. A total of 78 patients were enrolled and first completed a course of CBTI over a six week period. They they were randomized to of of the two tapering conditions or to a control (CTRL) condition in which their medication was not tapered. After the 20 week tapering period the study blind was eliminated and those in the CTRL condition were offered an open label tapering period. All patients were assessed for hypnotic use at the end of their respective tapering periods and then again 3 months later. Study key outcome measures included hypnotic discontinuation rates, nights per week hypnotics were used and weekly diazepam dose equivalents of hypnotics used. This line of research should inform clinical practice by helping to refine guidelines for tapering controlled substance hypnotic medications.

DETAILED DESCRIPTION:
Treatment seeking insomnia sufferers most often present in primary care venues where the first and usually only treatment is a prescription for a sedative hypnotic, typically a benzodiazepine or newer benzodiazepine receptor agonist, For some patients, short term or intermittent use provides satisfactory insomnia relief. However, more than 65 percent of individuals who are prescribed hypnotics use them for more than a year, and over 30 percent remain on these agents for more than five years. Whereas some patients may appreciate partial or full relief of insomnia symptoms with ongoing hypnotic use, continuous long-term use of these agents may not represent optimal therapy. Many insomnia patients who participate in non drug insomnia therapy such as as cognitive behavioral insomnia therapy or CBTI achieve sustained insomnia remission lon after a time limited course of treatment. However it is difficult for most long term hypnotic users to convert to a self management approach. Intervention that combine CBTI with a supervised medication tapering or SMT have shown the greatest promise for achieving this outcome, but almost 50 percent of patients who receive this treatment either fail to discontinue hypnotics or resume them over time. Previous research provides only rudimentary understanding of how to help long term hypnotic users discontinue their sleep aids and successfully manage their insomnia with CBTI techniques. This R34 gathered key pilot data to address these limitations. Specifically this project compared the currently recommended tapering pace which is a 25 percent dose reduction every two weeks with a slower 10 percent dose reduction every two weeks. The study also conducted all tapering in double blinded fashion. A total of 78 patients were enrolled and first completed a course of CBTI over a six week period. They they were randomized to of of the two tapering conditions or to a control CTRL condition in which their medication was not tapered. After the 20 week tapering period the study blind was eliminated and those in the CTRL condition were offered an open label tapering period. All patients were assessed for hypnotic use at the end of their respective tapering periods and then again 3 months later. Study key outcome measures included hypnotic discontinuation rates, nights per week hypnotics were used and weekly diazepam dose equivalents of hypnotics used. This line of research should inform clinical practice by helping to refine guidelines for tapering controlled substance hypnotic medications.

ELIGIBILITY:
Inclusion Criteria:

1. be currently using one or more BZD or newer BzRA hypnotics at bedtime for insomnia management;
2. have been using one or more such agents at least 5 nights per week for at least the past 12 months;
3. express interest in discontinuing hypnotic use and learning to manage their insomnia without medications;
4. report one or more failed attempts to discontinue hypnotic use in the past;
5. provide written consent to participate.
6. have an insomnia severity index score > 10 indicating at least mild insomnia symptoms without sleep medication

Exclusion Criteria:

1. an untreated unstable, or "in-treatment" psychiatric disorder (e.g., major depression in psychotherapy or on a medication regimen that has been changed within the past 2 months)
2. a lifetime diagnosis of any psychotic or bipolar disorder
3. an imminent risk for suicide
4. evidence of alcohol or drug abuse (other than hypnotics) within the past year, since such abuse patterns suggest specialized substance abuse treatment may be indicated
5. unstable or terminal physical illness (e.g., cancer), neurological degenerative disease (e.g., dementia) or sleep disruptive medical condition (e.g. chronic pain)
6. current use of medications known to cause insomnia (e.g., corticosteroids)
7. a history or screening evidence of restless legs syndrome, circadian rhythm sleep disorder (e.g., delayed sleep phase syndrome), sleep apnea (AHI > 5), or periodic limb movement disorder (PLM index > 15)
8. habitual bedtimes later than 2:00 AM or rising times later than 10:00 AM; (i) consuming > 2 alcoholic beverages per day at least 5 times per week
9. pregnant women or mothers with care-taking responsibilities for infants due to the sleep-disruption caused by such circumstances.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Participant Dropout Rate As Assessed By Analysis of Participant Register | 20-week tapering phase
  Measurement will be taken by analysis of participant register of the proportion of participants in each tapering group who drop out before the end of the 20-week tapering period.
Hypnotic Discontinuation Rate As Assessed By Analysis of Study Pharmaceutical Records | 20-week tapering phase
  Measurement will be taken by analysis of study pharmaceutical records of the proportion of participants in each tapering group who achieve full withdrawal of their hypnotic medication at or before the end of the tapering protocol.

SECONDARY OUTCOMES:
Hypnotic Relapse Rate As Assessed by Analysis of Participant Reports | Three-month follow-up phase
  Measurement will be taken by analysis of participant reports of the proportion of participants in each tapering group who achieve medication abstinence but subsequently return to hypnotic use by the 3-month follow-up visit.
Time to Drop Out of the Tapering Protocol As Assessed by Analysis of Participant Register | 20-week tapering phase
  Measurement will be taken by analysis of participant register and drop out dates of the time between the beginning of the 20-week and the effective date of participant drop out.
Absolute Change/Reduction in Diazepam Equivalents of Medication Being Used Nightly As Assessed by Study Pharmaceutical Records | 20-week tapering phase and three-month follow-up phase
  Measurement will be taken by analysis of study pharmaceutical records of the absolute change or reduction in diazepam equivalents of medication being used nightly by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jack D Edinger, Ph.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Archives. All data related to the clinical trial will be placed in the public domain in a time frame consistent with NIMH policies. Primary datasets will be made available via CDROM. These datasets will not include any personal identification related to participants or clinical sites beyond the usual numerical keys. Variable dictionaries, detailing variable description, format, value domain and labels, will be produced. Raw data will be exported in comma-separated format, to be readable by all major statistical software. Archives will also include data collection instructions and scoring algorithms for inventories. All reading material will be archived in PDF format.

REFERENCES:
- [Derived] Edinger JD, Wamboldt FS, Johnson RL, Simmons B, Tsai S, Morin CM, Holm KE. Adherence to behavioral recommendations of cognitive behavioral therapy for insomnia predicts medication use after a structured medication taper. J Clin Sleep Med. 2023 Aug 1;19(8):1495-1503. doi: 10.5664/jcsm.10616. PMID 37086054